CLINICAL TRIAL: NCT05815446
Title: Diagnostic Accuracy of Non-Contrast Computed Tomography in Correlation With Ultrasound in Detecting Acute Appendicitis in Adults
Brief Title: Non Contrast CT in Acute Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Omar Mohamed Ali, Principal Investigator, Assiut University
Other Study IDs: CT in acute appendicitis
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT — NON CONTASR COMPUTED TOMOGRAPHY

SUMMARY:
To evaluate Diagnostic accuracy of Non-contrast CT in correlation with ultrasound in diagnosis of acute appendicitis in adults

DETAILED DESCRIPTION:
Acute appendicitis is a prevalent cause of abdominal pain, with an estimated lifetime risk of 7 to 9%.[1] Diagnosing appendicitis on CT has a sensitivity and specificity of 87% and 76%, respectively. Classically, diagnosis of acute appendicitis is by identifying an enlarged appendix (greater than 6 mm in diameter) .

Some studies suggest using a cut-off value of over 7 mm to improve the prognostic capability of CT.

On the other hand, appendicitis is regularly diagnosed using radiology studies. In fact, imaging is often the deciding factor between operative and non-operative management. Though the diagnosis can be clinical following a thorough history and physical, imaging is regularly employed to confirm the diagnosis in question. The most commonly used radiographic study is the CT scan, given its speed, sensitivity, and specificity. US is also relatively useful modality to diagnose acute appendicitis, it has its limitations. Ultrasound is highly operator dependent and tends to work best on individuals with less fat and muscle content in their abdomen (i.e., children). Currently, the negative appendectomy is less than 12% in men but can be up to 33% in women; accurate imaging studies could reduce the number of unnecessary surgeries performed on patients. It is, therefore, essential to know which study will provide the clinician with the most accurate information for their specific clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (male or female) with clinical suspicion of acute appendicitis .

Exclusion Criteria:

* pregnant ladies and patients with history of appendectomy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be applied upon all patient referred from the emergency ward with clinical suspicious of acute appendicitis during the period from April 2023 to December 2023. Patients should fulfill the following criteria.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of non contrast CT in correlation with ultrasound in acute appendicitis . | baseline
  Diagnostic Accuracy of Non-Contrast Computed Tomography in Correlation with Ultrasound in Detecting Acute Appendicitis in Adults.

REFERENCES:
- [Background] Cohen CI. A case report: periodontal surgery in Parkinsonism utilizing intravenous sedation. N Y State Dent J. 1978 Jan;44(1):19. No abstract available. PMID 271274
- [Background] Drazen JM. Asthma therapy with agents preventing leukotriene synthesis or action. Proc Assoc Am Physicians. 1999 Nov-Dec;111(6):547-59. doi: 10.1046/j.1525-1381.1999.t01-1-99242.x. PMID 10591083